CLINICAL TRIAL: NCT04093167
Title: A Biomarker-Directed, Multi-Centre Phase II/III Study of CTDNA Response Adaptive Immuno-Chemotherapy in Non-Small Cell Lung Cancer
Brief Title: Study of CTDNA Response Adaptive Immuno-Chemotherapy in NSCLC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Cancer Research Institute, New York City (Other); Personal Genome Diagnostics (Industry); Mark Foundation for Cancer Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR36; CRI-CCTG-002 (Other: CRI)
Record Dates: First submitted 2019-09-12; First posted 2019-09-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pembrolizumab alone (Active Comparator)
  Interventions: Drug: Pembrolizumab
- Pembrolizumab + standard platinum-based chemotherapy (Experimental)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Per current Product Monograph/U.S. Drug Label and/or local guidelines.

SUMMARY:
BR36 will evaluate the potential clinical benefit of tailoring immunotherapy treatment based on ctDNA molecular response in non-small cell lung cancer.

DETAILED DESCRIPTION:
BR36 is an international multi-centre, open-label, biomarker-directed, phase II/III trial of ctDNA response adaptive immuno-chemotherapy in patients with immune checkpoint and chemotherapy naïve metastatic non-small cell lung cancer with ≥50% PD-L1 TPS expression. This trial will test if adding chemotherapy to pembrolizumab for patients with persistent ctDNA on Liquid Biopsy drawn at 6 weeks of treatment will result in better progression-free and overall survival compared to patients who remain on pembrolizumab therapy until clinical progression with subsequent change in standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic NSCLC. Patients with stage III disease are eligible if they are not candidates for surgical resection or definitive chemoradiation. Patients with Large Cell Neuroendocrine Carcinoma (LCNEC) are not eligible.
* Confirmed EGFR and ALK mutation-negative disease based on testing consistent with local guidelines.
* Patients must have a PD-L1 test result from a certified laboratory indicating PD-L1 expression Tumour Proportion Score (TPS) ≥ 50%. Patients with lower PD-L1 TPS scores treated with single agent pembrolizumab consistent with local guidelines and regulatory approvals may be eligible following discussion with CCTG.
* Patients are to be registered prior to starting immunotherapy. Screening ctDNA is to be drawn following registration prior to starting immunotherapy and after not more than 2 cycles of the 200mg or 2mg/kg IV Q3W dose/schedule of pembrolizumab, or at least and not more than 1 cycle of 400mg or 4mg/kg IV Q6W dose/schedule of pembrolizumab as first-line systemic immunotherapy for advanced metastatic NSCLC at the time of. Eligible patients with detectable ctDNA at 6 weeks may proceed to enrollment and randomization.
* Prior chemotherapy or immunotherapy for non-metastatic disease (e.g. adjuvant and or neoadjuvant therapy) is allowed if at least 6 months have elapsed between the completion of prior therapy and start of pembrolizumab as first-line treatment for metastatic disease. Local therapy, e.g. palliative extra-cranial radiation, is allowed as long as a period of 2 weeks has passed since completion and screening as ctDNA levels may be altered by radiotherapy. There is no requirement for delay for patients who have received brain radiation.
* Patients must have recovered to ≤ grade 1 from all reversible toxicity related to prior systemic or radiation therapy.
* Previous major surgery is permitted provided that surgery occurred at least 14 days prior to screening of ctDNA and 28 days prior to patient enrollment and that wound healing has occurred.
* Eligible and suitable to receive continued treatment with pembrolizumab OR the addition of chemotherapy to pembrolizumab at the time of registration and again at the time of enrollment and randomization. Patients should be clinically stable without evidence of clinical progression or symptomatic deterioration that requires change in cancer treatment. Reimbursement of pembrolizumab may not be uniform across all sites. In the event that the site/investigator is unable to provide access to the drug, the patient will not be eligible for this trial.
* Must be ≥ 18 years of age.
* ECOG performance status 0-2.
* Clinically and/or radiologically documented and evaluable disease. Measurable disease as defined by RECIST is not required.
* Imaging investigations including CT of the chest, abdomen and pelvis and MRI/CT of the brain (if known brain metastases) or other scans as necessary to document all sites of disease must be done within 14 days prior to randomization to ensure patients do not have clinical progression requiring change in systemic treatment. Patients must have non-progression of disease to be randomized. Patients who are clinically stable with PD such that in the opinion of the investigator they could continue with single agent immunotherapy may be eligible for enrollment and randomization following discussion with CCTG.
* Patients must have RECIST non-PD or clinically stable PD documented prior to enrollment that can continue on IO therapy if randomized to that arm.
* Detectable ctDNA on screening at 6 weeks is required for subsequent enrollment and randomization.
* Adequate hematology and organ function to continue immunotherapy or receive standard platinum combination therapy (must be done prior to registration for ctDNA testing) and prior to enrollment and randomization).

  * White Blood Cells ≥ 2.0 x 10^9/L (2000/μL)
  * Absolute neutrophils ≥ 1.5 x 10^9/L (1500/μL)
  * Platelets ≥ 100 x 10^9/L (100 x 10^3/μL)
  * Bilirubin ≤ 1.5 x ULN (upper limit of normal)*
  * AST and/or ALT ≤ 3 x ULN, < 5 x ULN for patients with liver metastases
  * Serum creatinine or Creatinine clearance ≤ 1.5 x ULN OR ≥ 40 mL/min
* Patients must consent to the provision of, and investigator must agree to submit, a representative archival formalin-fixed paraffin block of tumour tissue for correlative analyses when tumour tissue is available.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to registration to the trial to document their willingness to the collection of liquid biopsy (blood) samples for ctDNA analysis by CLIA central laboratory and for correlative analysis by a research central laboratory, and to subsequent enrollment and randomization to continued pembrolizumab or the addition of chemotherapy to pembrolizumab if ctDNA is detected.
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients enrolled on this trial will be available for complete documentation of the treatment, adverse events, collection of blood samples, response assessments and follow-up. Patients must agree to return to their primary care facility for response assessments as well as any adverse events which may occur through the course of the trial.
* In accordance with CCTG policy, protocol treatment is to begin within 5 working days of patient randomization.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method during protocol treatment and for at least 6 months after the last dose of the protocol treatment. Participants of childbearing potential will have a pregnancy test to determine eligibility as part of the Pre-Study Evaluation. Male participants with partners of childbearing potential must agree to use condoms (with spermicide, if available) in combination with an additional highly effective contraceptive method used by their partner, during treatment period and for at least 6 months after the last dose of the investigational product.

Exclusion Criteria:

* Patients with a prior malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the protocol treatment regimens are eligible for this trial.
* Patients with symptomatic central nervous system (CNS) metastases and/or CNS metastases requiring immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone equivalents). Patients with known central nervous system metastases who are asymptomatic and on a stable dose of corticosteroids ≤ 10 mg/day prednisone equivalents are eligible.
* Patients who are not suitable candidates for treatment with pembrolizumab as a single agent or in combination with standard platinum combination chemotherapy according to the current guidance/indications described in the Product Monograph (Canada) or Drug Label (U.S.) and practice guidelines including but not limited to patients with active infection, autoimmune disease, conditions that require systemic immunosuppressive therapy (such as transplant patients) and patients with a history of severe immune-mediated adverse reactions, or known hypersensitivity to pembrolizumab or its components. Patients with pre-existing conditions such as colitis, hepatic impairment, respiratory or endocrine disorders (such as hypo or hyperthyroidism or diabetes mellitus), can be considered for enrollment to this study provided pembrolizumab is administered with caution and patients are closely monitored. Patients should not have contraindications to platinum combination chemotherapy.
* History of significant neurologic or psychiatric disorder that would impair the ability to obtain consent or limit compliance with study requirements.
* Concurrent treatment with other anti-cancer therapy or other investigational anti-cancer agents
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Concordance rate between molecular response and radiologic response | 18 months
  Molecular response will be assessed by measuring changes in ctDNA levels in plasma
Stage 2: Phase II Progression-Free Survival (PFS) | 3 years
Stage 2: Phase III Overall Survival | 3 years

SECONDARY OUTCOMES:
Stage 1: Time to molecular response | 18 months
Stage 1: Correlate molecular response to RECIST response based on changes in ctDNA levels | 18 months
Stage 1: Correlate molecular response to progression-free survival based on changes in ctDNA levels | 18 months
Stage 1: Correlate molecular response to overall survival based on changes in ctDNA levels | 18 months
Stage 1: Explore the degree of ctDNA reduction with clinical outcomes assessed by measuring changes in ctDNA levels in plasma | 18 months
Stage 2: Phase II - Feasibility defined as screening success greater than 30% of patients screened have persistent ctDNA post 6 weeks of pembrolizumab | 3 years
Stage 2: Phase II - Feasibility defined as accrual reaching 50% of project accrual by month 18 post randomization | 3 years
Stage 2: Phase II - Feasibility defined as acceptance of randomization defined as >/= 80% of consenting patients accept randomization | 3 years
Stage 2: Phase II - clinical efficacy endpoints of best overall response rate post randomization | 3 years
Stage 2: Phase II - Number and severity of adverse events assessed by CTCAE v5 | 3 years
Stage 2: Phase III - Clinical efficacy endpoints of best overall RECIST response rate post-randomization | 3 years
Stage 2: Phase III - Clinical efficacy endpoints of response duration | 3 years
Stage 2: Phase III - Clinical efficacy endpoints of progression-free survival | 3 years
Stage 2: Phase III - Number and severity of adverse events assessed by CTCAE v5 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Valsamo Anagnostou, Study Chair — Johns Hopkins University; Sara Moore, Study Chair — Ottawa Hospital Research Institute
Locations (6):
- The Sidney Kimmel Comprehensive Cancer Centre, Baltimore, Maryland, United States
- Canada (5):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anagnostou V, Ho C, Nicholas G, Juergens RA, Sacher A, Fung AS, Wheatley-Price P, Laurie SA, Levy B, Brahmer JR, Balan A, Niknafs N, Avrutin E, Zhu L, Sausen M, Bradbury PA, O'Donnell-Tormey J, Gaudreau PO, Ding K, Dancey J. ctDNA response after pembrolizumab in non-small cell lung cancer: phase 2 adaptive trial results. Nat Med. 2023 Oct;29(10):2559-2569. doi: 10.1038/s41591-023-02598-9. Epub 2023 Oct 9. PMID 37814061